CLINICAL TRIAL: NCT07004972
Title: A Phase 4, Single-Arm, Open-Label Study to Evaluate Safety, Tolerability, and Efficacy of Mavacamten in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy in India
Brief Title: A Study of Mavacamten in Adults With Obstructive Hypertrophic Cardiomyopathy in India (ROVER)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV027-1146
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mavacamten (Experimental)
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
  Other Names: BMS-986427

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of mavacamten in adults with obstructive hypertrophic cardiomyopathy in India.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with obstructive hypertrophic cardiomyopathy (HCM) consistent with current American College of Cardiology Foundation/American Heart Association and European Society of Cardiology guidelines.
* Has unexplained LV hypertrophy with nondilated ventricular chambers in the absence of other cardiac (ie, hypertension, aortic stenosis) or systemic disease and with maximal LV wall thickness ≥ 15 mm (or ≥ 13 mm with positive family history of hypertrophic cardiomyopathy).
* Has LVOT (Valsalva left ventricular outflow tract) peak gradient ≥ 50 mmHg during screening as assessed by TTE at rest, Valsalva maneuver, or post exercise LVOT peak gradient.
* Has LVOT peak gradient with Valsalva at screening TTE of ≥ 30 mmHg.
* Has adequate acoustic windows to enable accurate TTEs.
* Has New York Heart Association (NYHA) Class II or III symptoms at screening.
* Body weight is greater than 45 kg at screening.
* Documentation of LVEF ≥ 55% at rest of screening TTE.

Exclusion Criteria

* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics obstructive hypertrophic cardiomyopathy, such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy.
* Has paroxysmal atrial fibrillation present per the investigator's evaluation of the participant's ECG at the time of screening.
* Has persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to screening and/or not adequately rate controlled within 6 months prior to screening. (Note: Participants with persistent or permanent atrial fibrillation who are anticoagulated and adequately rate-controlled are allowed).
* Has a history of syncope with exercise within 6 months prior to screening.
* History of sustained ventricular tachyarrhythmia (> 30 seconds) within 6 months prior to screening.
* Has documented obstructive coronary artery disease (> 70% stenosis in one or more epicardial coronary arteries) or history of myocardial infarction.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious Treatment Emergent Adverse Events (TEAEs) | Up to Week 48

SECONDARY OUTCOMES:
Number of participants with major adverse cardiac events | Up to Week 48
  Major adverse cardiac events includes cardiovascular [CV] death, non-fatal stroke, nonfatal myocardial infarction and hospitalization for heart failure
Number of participants with CV hospitalization | Up to Week 48
Number of participants with heart failure (HF) events | Up to Week 48
  HF includes HF related hospitalizations and urgent emergency room [ER]/outpatient visits
Number of participants with atrial fibrillation/flutter | Up to Weeks 48
Number of participants with syncope | Up to Week 48
Number of participants with left ventricular ejection fraction (LVEF) < 50% | Up to Week 30
Number of participants with left ventricular ejection fraction (LVEF) < 45% | Up to Week 30
Number of participants with left ventricular ejection fraction (LVEF) < 40% | Up to Week 30
Number of participants with left ventricular ejection fraction (LVEF) < 30% | Up to Week 30
Number of participants with non-serious AEs | Up to Week 48
Change from baseline to Week 30 in Valsalva left ventricular outflow tract (LVOT) peak gradient | Up to Week 30
Change from baseline to Week 30 in resting LVOT peak gradient | Up to Week 30
Change from baseline to Week 30 in hs-troponin-I | Up to Week 30
Change from baseline to Week 30 in N-terminal pro b-type natriuretic peptide (NT-proBNP) | Up to Week 30
Proportion of participants with at least 1 class improvement in New York Heart Association (NYHA) functional class from baseline to Week 30 | Up to Week 30
  The New York Heart Association (NYHA) functional classification of heart failure assigns participants to 1 of 4 categories based on the participant's symptoms. Heart failure classification will be assessed by the Investigator at specified timepoints in the study. NYHA class at Week 30 will be compared to baseline and the proportion of participants with an improvement of at least one class will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- India (29):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Marengo CIMS Hospital, Ahmedabad, Gujarat
  - Unicare Heart Institute (A division of Unique Hospital), Surat, Gujarat
  - Medanta Heart Institute, Gurgaon, Haryana
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi, Karnataka
  - Omega Hospital, Mangalore, Karnataka
  - Amrita Hospital, Ernākulam, Kerala
  - Caritas Hospital, Kottayam, Kerala
  - ORIION Citicare Superspeciality Hospital, Aurangabad, Maharashtra
  - King Edward Memorial Hospital & Seth Gordhandas Sunderdas Medical College, Mumbai, Maharashtra
  - Local Institution - 0025, Mumbai, Maharashtra
  - Central India cardiology hospital and Research Ins, Nagpur, Maharashtra
  - Viveka Hospital, Nagpur, Maharashtra
  - All India Institute of Medical Sciences ( AIIMS ) - Nagpur, Nagpur, Maharashtra
  - Local Institution - 0024, Nagpur, Maharashtra
  - KEM Hospital Research Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0021, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0016, Bhubaneswar, Odisha
  - Local Institution - 0018, Cuttack, Odisha
  - Local Institution - 0015, Ludhiana, Punjab
  - Sardar Patel Medical College And Assoc. Group Of Hospitals, Bikaner, Rajasthan
  - Tamil Nadu Government Multi-Super-Specialty Hospital, Chennai, Tamil Nadu
  - Jawaharlal Nehru Medical College, Aligarh, Uttar Pradesh
  - Local Institution - 0022, Aligarh, Uttar Pradesh
  - Laxmipat Singhania Institute of Cardiology, Kanpur, Uttar Pradesh
  - Institute of Post Graduate Medical Education and Research (IPGMER) and SSKM Hospital, Kolkata, West Bengal
  - Local Institution - 0009, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html